CLINICAL TRIAL: NCT01005992
Title: Fractional Photothermolysis for the Treatment of Burn Scars
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Clinica las Condes, Chile (Other)
Collaborators: Corporacion de ayuda al niño quemado (COANIQUEM) (Unknown); Solta Medical (Industry)
Responsible Party: Rodrigo Schwartz M.D., Clinica Las Condes
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CLCCQFQ-1
Record Dates: First submitted 2009-10-30; First posted 2009-11-02 (Estimated); Last update posted 2009-11-02 (Estimated); Status verified 2009-10

CONDITIONS: Scar
Keywords: Scars secondary to injuries to tissues caused by contact with physical (heat, electricity) o chemical agent.
MeSH Terms: conditions — Cicatrix

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Laser treated scar (Experimental): The standard treated scar arm consists of a similar lesion in an equivalent location in the same patient or the half of a lesion that is suitable to be divided (size at least 4% body surface area). This arm will be managed only with standard burn treatment modalities.
  Interventions: Procedure: Fractional laser treatment
- Standard scar management (Active Comparator): The standard scar management arm consists of a similar lesion in an equivalent location in the same patient or the half of a lesion that is suitable to be divided (size at least 4% body surface area). This arm will be managed only with standard burn treatment modalities.
  Interventions: Procedure: Standard scar management

INTERVENTIONS:
Procedure: Fractional laser treatment — A complete treatment will consist in four laser sessions with a second-generation erbium-doped 1,550-nm fractional photothermolysis laser (Fraxel SR laser, Reliant Technologies Inc at 1-month intervals. Treatment will be delivered with a 15-mm tip and concomitant air-cooling system (Zimmer MedizinSystems, Irvine, CA). Fluence and treatment level will be registered on every session and will be adjusted according to patient tolerance.
  Arms: Laser treated scar
Procedure: Standard scar management — The standard treated scar arm consists of a similar lesion in an equivalent location in the same patient or the half of a lesion that is suitable to be divided (size at least 4% body surface area). This arm will be managed only with standard burn treatment modalities.
  Arms: Standard scar management

SUMMARY:
The aim of our study is to determine the effect of fractional photothermolysis laser in the treatment of burn scars.

DETAILED DESCRIPTION:
One of the main problems in the management of burned patients is the treatment of post-burn scarring. Frequently this scars cover large areas, tend to retract, present pigmentary changes and are disfiguring, producing significant life quality impairment.

Unfortunately, there are very few therapeutic options for treating these scars, which can be secondary to reconstructive surgery or after spontaneous healing. In the last decades most reports in scar treatment have included, pressure garments, chemical peeling, dermabrasion, ablative and non-ablative laser therapy and surgery with varying degrees of success. There is only one report treating burn scars with fractional laser, with good results.

The aim of our study is to determine the effect of of a second-generation erbium-doped 1,550-nm fractional photothermolysis laser (Fraxel SR laser, Reliant Technologies Inc.) in the treatment of burn scars.

ELIGIBILITY:
Inclusion Criteria:

* Burn scars should be located on the anterior thorax or abdomen with at least 4 months of evolution.
* The scar should be slightly elevated, with erythema and with no signs of keloid formation.
* Maximum scar dimension: 0.2 - 1% body surface area.
* Acceptance of informed consent for laser treatment.

Exclusion Criteria:

* Previous non-surgical treatment (i.e. dermabrasion, laser, peelings, bleaching agent. etc).
* Previous surgical treatment (i.e. graft)

Ages: 6 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 10 (Estimated)
Dates: Start 2009-11; Primary Completion 2010-04 (Estimated)

PRIMARY OUTCOMES:
Evidence of improvement in color and texture of burn scars, using digital colorimeter and digital photography. | 5 months
Adverse effects: pain, erythema, edema, hypopigmentation, hyperpigmentation, hypertrophic scar and keloid formation | 5 months

SECONDARY OUTCOMES:
Change in surface area and perimeter of burn scar | 5 months
Tissue pliability, elevation and flexibility with a digital piedemeter | 5 months
Change in collagen fiber organization and blood vessel density with a reflectance laser confocal microscope. | 5 months

CONTACTS AND LOCATIONS:
Overall Officials: Rodrigo J Schwartz, MD, Principal Investigator — Clinica Las Condes
Locations (1):
- Clinica Las Condes, Santiago, RM, Chile

REFERENCES:
- [Background] Chrastil B, Glaich AS, Goldberg LH, Friedman PM. Second-generation 1,550-nm fractional photothermolysis for the treatment of acne scars. Dermatol Surg. 2008 Oct;34(10):1327-32. doi: 10.1111/j.1524-4725.2008.34284.x. PMID 19040687
- [Background] Glaich AS, Rahman Z, Goldberg LH, Friedman PM. Fractional resurfacing for the treatment of hypopigmented scars: a pilot study. Dermatol Surg. 2007 Mar;33(3):289-94; discussion 293-4. doi: 10.1111/j.1524-4725.2007.33058.x. PMID 17338685
- [Background] Haedersdal M. Fractional ablative CO(2) laser resurfacing improves a thermal burn scar. J Eur Acad Dermatol Venereol. 2009 Nov;23(11):1340-1. doi: 10.1111/j.1468-3083.2009.03215.x. Epub 2009 Mar 4. No abstract available. PMID 19309424
- [Background] Haedersdal M, Moreau KE, Beyer DM, Nymann P, Alsbjorn B. Fractional nonablative 1540 nm laser resurfacing for thermal burn scars: a randomized controlled trial. Lasers Surg Med. 2009 Mar;41(3):189-95. doi: 10.1002/lsm.20756. PMID 19291747
- [Background] Waibel J, Beer K. Fractional laser resurfacing for thermal burns. J Drugs Dermatol. 2008 Jan;7(1):59-61. PMID 18246699
- [Background] Waibel J, Beer K. Ablative fractional laser resurfacing for the treatment of a third-degree burn. J Drugs Dermatol. 2009 Mar;8(3):294-7. PMID 19271380